CLINICAL TRIAL: NCT06384625
Title: Developing and Evaluating an Indoor Air Pollution Intervention Among Cardiovascular Patients: the AIRWISE Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Montana (Other)
Collaborators: Providence Heart Institute (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 361378
Record Dates: First submitted 2024-04-11; First posted 2024-04-25 (Actual); Last update posted 2025-11-10 (Actual); Status verified 2025-06

CONDITIONS: Coronary Heart Disease; Cardiovascular Diseases; Environmental Exposure
MeSH Terms: conditions — Coronary Disease; Cardiovascular Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Air pollution intervention implementation (Other): AIRWISE intervention implementation
  Interventions: Other: AIRWISE

INTERVENTIONS:
Other: AIRWISE — AIRWISE (Air Improvement and Real-time Monitoring for Wellness through Interactive Strategies and Education) utilizes personal air cleaners (PACs) to filter indoor air, while enhanced aspects focus on improving compliance to PAC use. Key components include low-cost sensors (PurpleAir, Inc, USA) that change color according to air quality index (AQI) and behavioral recommendations that correspond to varying AQI levels.

SUMMARY:
This pilot study (n=20) is a prospective evaluation of the implementation of an indoor air pollution intervention among adults 55 years of age or older. The intervention, called Air Improvement and Real-time Monitoring for Wellness through Interactive Strategies and Education (AIRWISE), is focused on improving indoor air quality through air filtration, education, and behavioral recommendations. All participants will receive the AIRWISE intervention with the objective of evaluating acceptance and use of the individual intervention components. This implementation study will inform the submission of a larger NIH proposal for a randomized trial. The central study hypothesis is that an intervention program with educational strategies and visual behavioral cues will increase knowledge and awareness of air pollution exposures among the participants and lead to improved intervention compliance.

ELIGIBILITY:
Inclusion Criteria:

* Adult of at least 55 years of age
* One primary residence (5+ days per week)
* Own a computer or electronic device (tablet or phone with web browser), and reliable internet connection or cell phone service (required to submit study surveys)
* Access to a working email address (required to submit study surveys)
* Electricity in the home (required to power the study equipment)

Exclusion Criteria:

* Current smoking of any kind (tobacco, cannabis, vape pens, cigars, etc.) or living in a household with someone who currently smokes
* Current use of stand-alone home high efficiency purified air (HEPA) filtration or PAC unit in the home
* Intention to move in the next 6 months
* Another person in the household is enrolled in this study (one person per household can enroll)
* Having any health condition that prevents the participants from having blood pressure measured using an upper-arm cuff: lymphedema, paresis or paralysis, arterial or venous lines/catheters, dialysis shunt, recent surgical wounds, or mastectomy

Min Age: 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2024-07-24 (Actual); Primary Completion 2025-11-05 (Actual); Study Completion 2025-11-05 (Actual)

PRIMARY OUTCOMES:
Evaluate the implementation of an indoor air pollution intervention. | 6 months
  As an implementation study, the investigators will administer the AIRWISE intervention to 20 adult participants (55+ years of age) and evaluate intervention fidelity, acceptance, and compliance over a 6-month period spanning the 2024 wildfire season. An important outcome measure is to understand how frequently participants use the primary intervention components that include personal air cleaners (PACs), an indoor air quality monitor that changes color based on air quality index, and educational materials. These 3 components will be evaluated via electronic surveys administered every 2 weeks over the course of the study. The investigators will use 7 Likert Scale (ordinal) questions to measure frequency of use for the intervention components. The 7 questions will be combined into a composite score of intervention use that ranges from 7 to 39, with higher scores indicating higher intervention use.

SECONDARY OUTCOMES:
Fine particulate matter (PM2.5) | 6 months
  Measure indoor PM2.5 concentrations among participant households during intervention evaluation.
Life's Essential 8 | 6 months
  The investigators will prospectively collect health measures to calculate a metric called Life's Essential 8 (LE8), a construct of cardiovascular health including blood pressure, lipids, glucose, body mass index, nicotine exposure, diet, physical activity, and sleep health. LE8 ranges from 0 to 100, with the score calculated as an unweighted average of the 8 component metric scores. Overall scores of 80 to 100 are considered high, 50 to 79 considered moderate, and 0 to 49 considered low. The investigators will then assess associations between the LE8 metric and indoor PM2.5 concentrations measured using the AIRWISE sensors. The hypothesis is that higher indoor PM2.5 concentrations over the course of the study will be associated with lower LE8 scores.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Montana, Missoula, Montana, United States

IPD SHARING:
Plan to Share IPD: No